CLINICAL TRIAL: NCT05918029
Title: Bone in CKD Alkali Response Pilot Trial (BICARb)
Brief Title: Bone in CKD Alkali Response (BICARb Pilot Trial)
Acronym: BICARb
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Columbia University (Other); University of Pittsburgh Medical Center (Other); University of Utah (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-14826; R01DK131811 (NIH)
Record Dates: First submitted 2023-06-02; First posted 2023-06-26 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Chronic Kidney Diseases; Bone Loss
Keywords: Chronic Kidney Disease; Bone strength; Fractures; Pediatrics; Metabolic acidosis
MeSH Terms: conditions — Renal Insufficiency, Chronic; Bone Diseases, Metabolic; Fractures, Bone; Acidosis | interventions — Potassium Citrate; Citric Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Potassium Citrate (Experimental): Potassium Citrate extended-release tablets 30 mEq twice daily. 1 mEq/kg/day divided into two doses for children to a maximum dose of 30 mEq twice daily.
  OR
  (for children who cannot take pills): Potassium citrate and citric acid for oral solution 1 mEq/kg/day divided into two doses to a maximum dose of 30 mEq twice daily
  Interventions: Drug: Potassium Citrate Extended Release Oral Tablet; Drug: Potassium Citrate and Citric Acid Oral Solution
- Placebo (Placebo Comparator): Placebo capsules identical to the active capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Potassium Citrate Extended Release Oral Tablet — Oral potassium citrate extended-release tablet
  Arms: Potassium Citrate
Other: Placebo — Placebo capsule identical to active ingredient
  Arms: Placebo
Drug: Potassium Citrate and Citric Acid Oral Solution — Oral potassium citrate and citric acid
  Arms: Potassium Citrate

SUMMARY:
The goal of this clinical trial is to test whether potassium citrate improves skeletal health in adults and children with chronic kidney disease. The main questions it aims to answer are:

* To evaluate effects of potassium citrate treatment on bone quality and strength.
* To evaluate mechanism(s) underlying the effects of potassium citrate on skeletal health.

Participants will be asked to:

* provide blood, urine and answer questions about health and diet three times during an 8 months period
* undergo advanced bone imaging with high resolution-peripheral quantitative CT scan twice during 8 months
* take study pills for 4-6 weeks at the beginning of the study to ensure safety
* take either potassium citrate or placebo for 6 months during the blinded portion of the study

As part of the study, there will be a run-in period followed by the placebo-controlled randomized clinical trial. Researchers will compare the bone imaging between the potassium citrate and the placebo groups at the end of the study.

DETAILED DESCRIPTION:
Chronic kidney disease is associated with bone loss and fractures in both children and adults, but bone protective therapies that are both proven and safe to use across the life-course in CKD are lacking. In this study, the investigators will conduct a pilot, double-blinded, randomized, placebo-controlled trial in 15 children and 88 adults evaluating the skeletal effects of potassium alkali therapy. These data will form the basis for a larger U01 proposal to determine the efficacy of potassium citrate on mitigating the effects of CKD on bone.

ELIGIBILITY:
Inclusion Criteria (Pediatric Inclusion):

* Children 5-17 years old
* Estimated eGFR >30 and <90 ml/min/1.73m2 by CKiD U25 equations
* Females of child-bearing potential must have had a menstrual period in the last month
* Levels of PTH and alkaline phosphatase within 2x normal range and phosphorus within the normal range for age (per local laboratory reference assay)
* 25-hydroxy Vitamin D ≥ 20 ng/mL
* Females of child-bearing potential must be willing to use one form of effective contraception over the course of the study
* Proficiency in English or Spanish
* For participants < 18 years, the participant and/or parent/guardian capable of providing informed consent and assent (assessed by the provider)

Inclusion Criteria (Adult Inclusion):

* Adults ≥ 18 years old
* Estimated eGFR >30 and <90 ml/min/1.73m2 by the new CKD-Epi without race
* Pre-menopausal women of childbearing age must have had a menstrual period in the last month
* Levels of PTH and alkaline phosphatase within 2x normal range and phosphorus up to 5.0 mg/dL (per local laboratory reference assay)
* Levels of 25-hydroxy Vitamin D ≥ 20 ng/mL
* Women of childbearing potential must be willing to use one form of effective contraception over the course of the study
* Proficiency in English or Spanish

Exclusion Criteria (Pediatric and Adult):

* Baseline potassium ≥ 5.5 mEq/L or prior history of hyperkalemia in the last 6 months (potassium > 5.5 mEq/L) or currently taking a potassium lowering agent
* Alkali therapy within the prior 12 months
* Baseline ECG with abnormalities associated with increased risk of arrythmia, excluding left ventricular hypertrophy
* Baseline serum bicarbonate levels < 17 or ≥ 30 mEq/L
* Serum calcium < 8.6 mg/dL, adjusted for serum albumin
* Significant comorbidity causing acid-base imbalance (e.g., active cancer requiring chemotherapy, chronic liver failure, moderate or severe chronic obstructive lung disease, New York Heart Association class 2 or greater congestive heart failure, obstructive sleep apnea requiring nightly continuous positive airway pressure, active glomerular disease requiring immunosuppressive therapy, intestinal malabsorption or celiac disease)
* Plans to relocate out of the area in the next 3 months
* Urine pH > 8 or history of nephrolithiasis
* Lower extremity amputations or non-ambulatory
* Metabolic bone disease not related to CKD (e.g., Paget's disease, primary hyperparathyroidism)
* Endocrinopathy: untreated hyper or hypothyroidism, Cushing's syndrome
* Medical diseases that can affect therapy (severe myocardial damage, acute dehydration, delayed gastric emptying, esophageal compression, or intestinal obstruction or stricture)
* Use of bisphosphonates, denosumab, teriparatide, abaloparatide, romosozumab, raloxifene, estrogen or testosterone replacement therapy, or an unstable dose of glucocorticoids within the 12-months prior to enrollment
* Previous bilateral wrist and tibia fractures
* Solid or liquid organ transplant
* On dialysis or with rapidly deteriorating kidney function or expectation for transplantation or initiation of dialysis in less than 3 months
* Pregnancy or breastfeeding
* Prisoners or institutionalized individuals
* Unwillingness to provide informed consent

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Change in Total volumetric bone mineral density (BMD) - Distal Radius | Baseline to 6 months
  Change in total volumetric BMD will be analyzed by high resolution peripheral quantitative computed tomography (HR-pQCT). The 6-month absolute and relative (percent) changes in Z-score in distal radius total volumetric BMD will summarized by study arm and analyzed for between group treatment changes.
Change in Total volumetric bone mineral density (BMD) - Tibia | Baseline to 6 months
  Change in total volumetric BMD will be analyzed by high resolution peripheral quantitative computed tomography (HR-pQCT). The 6-month absolute and relative (percent) changes in Z-score in tibia total volumetric BMD will summarized by study arm and analyzed for between group treatment changes.

SECONDARY OUTCOMES:
Change in 24-hour Urine Net Acid Excretion (NAE) | Baseline to 6 months
  Change in 24-hour urinary NAE from baseline will be assessed by analyzing samples obtained from 24-hour timed urine collections using laboratory titration methods. Results will be quantified and summarized by study arm using basic descriptive statistics and subsequently analyzed for between group treatment changes. Standard urinary NAE values vary but can range from 250-750 mg/24 hours (1.48 to 4.43 mmol/24 hours).
Change in Parathyroid Hormone (PTH) levels | Baseline to 6 months
  Change in circulating PTH concentration from baseline will be assessed by the collection of blood samples via venipuncture and analysis for circulating PTH by an immunoassay. Results will be summarized by study arm using basic descriptive statistics and subsequently statistically analyzed for between group changes. Standard PTH reference ranges can vary but are generally between 10-65 pg/mL in plasma.
Change in circulating biomarkers of bone resorption | Baseline to 6 months
  Change in circulating biomarkers of bone resorption from baseline will be assessed following the collection of blood samples via venipuncture and subsequent analysis for circulating C-terminal telopeptides of type I collagen using a cross-linking telopeptide of type I collagen (CTX blood test) assay. C-terminal telopeptides can be used as a biomarker to measure bone resorption and turnover. Elevated levels of C-terminal telopeptide can be indicative of increased bone resorption. While standard reference ranges for C-terminal telopeptide can vary, for premenopausal women ranges are typically 40-465 pg/mL in serum and 19-83 ug/L in plasma.
Change in circulating biomarkers of bone formation | Baseline to 6 months
  Change in circulating biomarker of bone formation from baseline will be assessed following the collection of blood samples via venipuncture and subsequent analysis for procollagen type-1 N-terminal propeptide (P1NP). A P1NP assay measures the amount of amino-terminal propeptide of type I procollagen in the serum and can be used as biomarker to measure the rate of bone formation. While reference ranges can vary by age, standard reference ranges in adult premenopausal women are 19-83 ug/L.

OTHER OUTCOMES:
Correlation of serum bicarbonate and urine NAE | 6 months
  Correlation coefficient will be determined between serum bicarbonate and urine net acid excretion. The correlation coefficient is a number between 0 and 1, with 0 being no correlation and 1 being perfect correlation.
Correlation of serum bicarbonate and bone quality | 6 months
  Correlation coefficient will be determined between serum bicarbonate and bone quality. The correlation coefficient is a number between 0 and 1, with 0 being no correlation and 1 being perfect correlation.
Correlation between urine net acid excretion and bone quality | 6 months
  Correlation coefficient will be determined between urine net acid excretion and bone quality. The correlation coefficient is a number between 0 and 1, with 0 being no correlation and 1 being perfect correlation.
Changes in bone alkaline phosphatase | 6 months
  Changes in bone alkaline phosphatase will be compared between the groups. Bone alkaline phosphatase is measured in IU/L. Higher values are indicative of higher bone turnover.
Changes in TRAP5b | 6 months
  Changes in TRAP5b compared between the groups. TRAP5b are measured in mIU/mL.
Changes in bone quality | 6 months
  Bone quality as measured by high resolution peripheral quantitative CT will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Reidy, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine, The Bronx, New York
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kilduff S, Brown DD, Melamed ML. Treating Metabolic Acidosis for CKD Progression? Need for Higher Quality Data. Clin J Am Soc Nephrol. 2025 Jan 1;20(1):147-149. doi: 10.2215/CJN.0000000632. Epub 2024 Nov 20. No abstract available. PMID 39665575